CLINICAL TRIAL: NCT05061095
Title: Understanding What Matters Most to Patients: Establishing the Validity of a Best-Worst Scaling Survey
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC 2136; U2CNR014637 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-29 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Neoplasms
Keywords: leukemia; lymphoma; myeloma; myelodysplastic syndrome; best-worst scaling survey
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment Surveys — Patients will complete surveys in three periods. An initial baseline survey, longitudinal assessments completed every 2 weeks over the course of the first three months on study (6 times maximum), and extended assessments that will happen every 3 months after the initial longitudinal period up to 2 years on the study (7 times maximum). Baseline questionnaire will collect demographic and background medical record information. Longitudinal assessments will consist of a BWS questionnaire (patients rate importance of 7 treatment goals), decisional conflict scales, EQ-5D-5L, distress thermometer, and items from PRO-CTCAE. Extended assessments will use same questionnaires as longitudinal assessments.
Other: Qualitative Interviews — Patients will participate in 2 interviews (1 initial interview, 1 follow up). These will be cognitive interviews focusing on establishing content validity for BWS questionnaire. Will establish patient understanding of questions asked in BWS, understanding of how preferences affect treatment decisions, expected outcomes, and feedback from patients on other potentially important attributes not included in BWS.

SUMMARY:
This study will evaluate the validity of using a survey to quantify patient preferences at the point-of-care and the potential effectiveness of the survey to improve goal-concordant care. The primary hypothesis is that by identifying the strength of patient preferences for outcomes with this survey clinicians will be able to improve goal-concordant care by aligning clinical recommendations with patients' preferences. This study will have 50 patients with newly diagnosed hematologic malignancy complete the survey throughout their disease course (up to 2 years) and conduct qualitative interviews with a subset (n = 20) of participants. The information obtained from these participants will be used to refine the survey. Interviews with oncologists and palliative care specialists (up to 10) will inform implementation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new diagnosis of one of the following hematologic malignancies: aggressive lymphoma, multiple myeloma, CLL, CML, AML, ALL, MDS EB1 or EB2
* Age≥60
* Ability to read, understand, and communicate fluently in English
* Ability to understand and comply with study procedures
* Willingness and ability to provide written informed consent

Exclusion Criteria:

* Dementia, altered mental status, or psychiatric condition that would prohibit the understanding or rendering of informed consent or participation in the discrete choice experiment.
* Significant medical conditions, as assessed by the investigators, that would substantially increase the burden on the patient to complete study assessments (such as multiorgan failure, respiratory failure, or other critical illness).

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants are older (≥60) patients with newly-diagnosed hematological malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Richardson, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson DR, Crossnohere NL, Seo J, Estey E, O'Donoghue B, Smith BD, Bridges JFP. Age at Diagnosis and Patient Preferences for Treatment Outcomes in AML: A Discrete Choice Experiment to Explore Meaningful Benefits. Cancer Epidemiol Biomarkers Prev. 2020 May;29(5):942-948. doi: 10.1158/1055-9965.EPI-19-1277. Epub 2020 Mar 4. PMID 32132149
- [Background] Richardson DR, Oakes AH, Crossnohere NL, Rathsmill G, Reinhart C, O'Donoghue B, Bridges JFP. Prioritizing the worries of AML patients: Quantifying patient experience using best-worst scaling. Psychooncology. 2021 Jul;30(7):1104-1111. doi: 10.1002/pon.5652. Epub 2021 Feb 27. PMID 33544421
- [Background] Seo J, Smith BD, Estey E, Voyard E, O' Donoghue B, Bridges JFP. Developing an instrument to assess patient preferences for benefits and risks of treating acute myeloid leukemia to promote patient-focused drug development. Curr Med Res Opin. 2018 Dec;34(12):2031-2039. doi: 10.1080/03007995.2018.1456414. Epub 2018 Apr 27. PMID 29565196
- [Background] Bridges JF, Oakes AH, Reinhart CA, Voyard E, O'Donoghue B. Developing and piloting an instrument to prioritize the worries of patients with acute myeloid leukemia. Patient Prefer Adherence. 2018 Apr 27;12:647-655. doi: 10.2147/PPA.S151752. eCollection 2018. PMID 29731612
- [Background] LeBlanc TW, Fish LJ, Bloom CT, El-Jawahri A, Davis DM, Locke SC, Steinhauser KE, Pollak KI. Patient experiences of acute myeloid leukemia: A qualitative study about diagnosis, illness understanding, and treatment decision-making. Psychooncology. 2017 Dec;26(12):2063-2068. doi: 10.1002/pon.4309. Epub 2016 Dec 19. PMID 27862591
- [Background] Loh KP, Abdallah M, Kadambi S, Wells M, Kumar AJ, Mendler JH, Liesveld JL, Wittink M, O'Dwyer K, Becker MW, McHugh C, Stock W, Majhail NS, Wildes TM, Duberstein P, Mohile SG, Klepin HD. Treatment decision-making in acute myeloid leukemia: a qualitative study of older adults and community oncologists. Leuk Lymphoma. 2021 Feb;62(2):387-398. doi: 10.1080/10428194.2020.1832662. Epub 2020 Oct 11. PMID 33040623
- [Background] Rood JAJ, Nauta IH, Witte BI, Stam F, van Zuuren FJ, Manenschijn A, Huijgens PC, Verdonck-de Leeuw IM, Zweegman S. Shared decision-making and providing information among newly diagnosed patients with hematological malignancies and their informal caregivers: Not "one-size-fits-all". Psychooncology. 2017 Dec;26(12):2040-2047. doi: 10.1002/pon.4414. Epub 2017 Apr 17. PMID 28264148
- [Background] El-Jawahri A, Nelson-Lowe M, VanDusen H, Traeger L, Abel GA, Greer JA, Fathi A, Steensma DP, LeBlanc TW, Li Z, DeAngelo D, Wadleigh M, Hobbs G, Foster J, Brunner A, Amrein P, Stone RM, Temel JS. Patient-Clinician Discordance in Perceptions of Treatment Risks and Benefits in Older Patients with Acute Myeloid Leukemia. Oncologist. 2019 Feb;24(2):247-254. doi: 10.1634/theoncologist.2018-0317. Epub 2018 Aug 23. PMID 30139841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 03/21/2022 through 06/29/2023 at one cancer center, in North Carolina. Subjects were enrolled in the study between 03/31/2022 through 06/29/2023.
Pre-assignment Details: A total of fifty-one participants consented and were eligible for the study, but twenty-seven of them started the study interventions.
Groups:
- All Participants: Participants who consented to participate.
Period: Overall Study
Arm/Group | All Participants
Started | 51
Enrolled and Registered | 27
Completed | 19
Not Completed | 32

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 71 [61 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 45
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 51
Primary diagnosis [Count of Participants; unit: Participants]
  Leukemia | 23
  Lymphoma | 22
  Multiple Myeloma | 2
  Blastic Plasmacytoid Dendritic Cell Neoplasm | 1
  Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Content Validity of Best-Worst Scaling (BWS) Survey
Description: Cognitive interviewing will be used to evaluate the content validity of using a BWS survey to quantify the preferences of older patients with hematologic malignancies at the point-of-care. BWS survey asks patients a series of questions where they choose one attribute as best and one as worst - the 7 included in this survey are maintaining usual activities, living longer, avoiding dependence on others, avoiding short-term side effects, avoiding long-term side effects, avoiding hospitalizations, and avoiding high out-of-pocket costs.
Time Frame: 3 months after treatment decision
Population: Participants with newly-diagnosed hematologic malignancies who completed cognitive interviews.
Measure: Count of Participants; unit: Participants
Groups:
- Qualitative Interviews: Participants (subset of the entire cohort) who completed cognitive interviews to establish the content validity of the BWS survey.
Arm/Group | Qualitative Interviews
Number analyzed (Participants) | 10
Participants
  Participants who were able to accurately define each attribute and reported no missing domains. | 10
  Participants who could not define attributes or reported missing domains. | 0

2. Secondary Outcome: Acceptability of Best-Worst Scaling (BWS) Survey to Patients
Description: Number of patients who respond with agree/strongly agree to "I found survey acceptable to clarify my preferences"
Time Frame: Up to 7 days after treatment decision
Population: Participants with newly-diagnosed hematologic malignancies who completed Best-Worst Scaling (BWS) survey.
Measure: Count of Participants; unit: Participants
Groups:
- Pilot Testing: Participants With Newly-diagnosed Hematologic Malignancies: Participants diagnosed participating in the questionnaire portion of the study.
Arm/Group | Pilot Testing: Participants With Newly-diagnosed Hematologic Malignancies
Number analyzed (Participants) | 19
Participants | 13

3. Secondary Outcome: Preliminary Efficiency of Best-Worst Scaling (BWS) Survey
Description: Number of patients who respond moderately effective/very affective to "how effective was the survey to help you and your doctor choose a treatment that was consistent with your goals?"
Time Frame: Up to 7 days after treatment decision
Population: Participants with newly-diagnosed hematologic malignancies who completed survey.
Measure: Count of Participants; unit: Participants
Groups:
- Pilot Testing:: Participants with newly-diagnosed hematologic malignancies who participated in the questionnaire portion of the study.
Arm/Group | Pilot Testing:
Number analyzed (Participants) | 19
Participants | 9

4. Secondary Outcome: Completion Rate Over Time
Description: The completion rate over time will be reported by the number of patients who complete the BWS survey at each time point, in 3 months intervals.
Time Frame: Up to 1 year
Population: Subjects signed the consent form
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 51
Participants
  consented | 51
  started BWS instrument at baseline | 27
  completed BWS instrument at baseline | 26
  completed study-associated surveys after their treatment encounter at least 1 time | 19
  completed study-associated surveys after their treatment encounter more than 1 time (median 8 times) | 16

ADVERSE EVENTS:
Time Frame: Not available. The protocol does not require adverse event assessment.
Description: The protocol does not require adverse event assessment. Adverse Event data was not collected.
Groups:
- All Participants: Participants who consented to participate and started to study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT05061095/Prot_SAP_000.pdf